CLINICAL TRIAL: NCT01503736
Title: A Randomized, Double-Blind, Placebo-Controlled, Multi-Center, Definitive Phase III Study of the Effects of Ferric Citrate on Serum Phosphate in Subjects With End Stage Renal Disease
Brief Title: A Randomized, Double-Blind, Placebo-Controlled Phase 3 Study of the Effects of Ferric Citrate in Subjects With End Stage Renal Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Panion & BF Biotech Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PNC00301
Record Dates: First submitted 2012-01-02; First posted 2012-01-04 (Estimated); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Hyperphosphatemia; End Stage Renal Disease; ESRD
Keywords: Kidney Diseases; Kidney Failure, Chronic; Hyperphosphatemia; Urologic Diseases; Renal Insufficiency, Chronic; Renal Insufficiency; Phosphorus Metabolism Disorders
MeSH Terms: conditions — Hyperphosphatemia; Kidney Failure, Chronic; Kidney Diseases; Urologic Diseases; Renal Insufficiency, Chronic; Renal Insufficiency; Phosphorus Metabolism Disorders | interventions — ferric citrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Placebo Comparator)
  Interventions: Drug: ferric citrate
- 4g/day (Experimental): Ferric Citrate for a total daily dose of 4g
  Interventions: Drug: ferric citrate
- 6g/day (Experimental): Ferric Citrate for a total daily dose of 6g
  Interventions: Drug: ferric citrate

INTERVENTIONS:
Drug: ferric citrate — 0g/day ferric citrate capsule, TID for 56 days
  Arms: Placebo
Drug: ferric citrate — 4g/day ferric citrate capsule, TID for 56 days
  Arms: 4g/day
Drug: ferric citrate — 6 g/day ferric citrate capsule, TID for 56 days
  Arms: 6g/day

SUMMARY:
The purpose of the study is to determine the effect and optimum dose and evaluate the safety of ferric citrate, administered three times daily (TID) immediately after meals for a total daily dose of 4 or 6 grams for 56 days, on serum phosphate (PO4) levels in subjects with end stage renal disease (ESRD).

ELIGIBILITY:
Inclusion Criteria:

* Age>18 years and has a diagnosis of ESRD
* On a three-times per week hemodialysis regimen
* On a stable dose of a phosphate-binding agent for at least one month prior to study entry.
* If on vitamin D supplementation or calcitriol, must be on a stable dose for at least one month prior to study entry.
* Hct >= 20%
* Serum Ca level of 8 mg/dL to 10.5 mg/dL

Exclusion Criteria:

* Is pregnant or lactating
* Clinically significant GI disorder
* Has tertiary hyperparathyroidism or is immediately post-operative from a parathyroidectomy (within the first 3 months post-op or the plasma Ca is <7 mg/dL)
* ferritin>800 ng/mL
* Unstable medical condition unsuitable for the study in the opinion of investigator
* Has been treated with an investigational agent within 30 days of enrollment
* Has a history of documented iron allergy or hemochromatosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 183 (Actual)
Dates: Start 2010-06; Primary Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Change in serum phosphorus at Day 56 as compared to baseline | Day 56

SECONDARY OUTCOMES:
Change in serum phosphorus at Day 28 as compared to baseline | Day 28
Change in Ca x P product at Day 56 compared to baseline | Day 56
Change in Ca x P product at Day 28 compared to baseline | Day 28
Cumulative drop out rate due to serum phosphorus concentration >9mg/dL at Day 56 | Day 56
Cumulative drop out rate due to serum Phosphorus concentration >9mg/dL at Day 28 | Day 28

CONTACTS AND LOCATIONS:
Locations (5):
- Taiwan (5):
  - Division of Nephrology, Department of Internal Medicine, Kaohsiung Chang-Gung Memorial Hospital, Kaohsiung City
  - Division of Nephrology, Keelung Chang Gung Memorial Hospital, Keelung
  - Division of Nephrology, Department of Internal Medicine, Far East Memorial Hospital, New Taipei City
  - Division of Nephrology, Department of Internal Medicine, Taichung Veterans General Hospital, Taichung
  - Division of Nephrology, Department of Internal Medicine, Shin Kong Wu Ho-Su Memorial Hospital, Taipei

REFERENCES:
- [Result] Lee CT, Wu IW, Chiang SS, Peng YS, Shu KH, Wu MJ, Wu MS. Effect of oral ferric citrate on serum phosphorus in hemodialysis patients: multicenter, randomized, double-blind, placebo-controlled study. J Nephrol. 2015 Feb;28(1):105-13. doi: 10.1007/s40620-014-0108-6. Epub 2014 May 20. PMID 24840781
- [Derived] Natale P, Green SC, Ruospo M, Craig JC, Vecchio M, Elder GJ, Strippoli GF. Phosphate binders for preventing and treating chronic kidney disease-mineral and bone disorder (CKD-MBD). Cochrane Database Syst Rev. 2025 Jun 27;6(6):CD006023. doi: 10.1002/14651858.CD006023.pub4. PMID 40576086